CLINICAL TRIAL: NCT04843605
Title: Impact of Systematic Screening for COPD in Tabacology Consultation
Brief Title: Systematic Screening for COPD in Tabacology Consultation
Acronym: DEBOTA
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC21.0036
Record Dates: First submitted 2021-04-09; First posted 2021-04-13 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
COPD is a very common disease, an estimated 3 million people are affected in France. Unfortunately, this pathology is under-diagnosed. Several reasons can be mentioned: the banality of the symptoms or the several comorbidities.

Screening faces a major difficulty: the realization of a spirometry. Various studies have shown the complexity of the implementation of mass screening in cities by mini-spirometry.

The COPD World Health Days allow this mass screening but without visibility on the actual entry into a care pathway.

The objective of this study is to assess the impact of systematic screening for COPD during a tabacology consultation

ELIGIBILITY:
Inclusion Criteria:

* Subjects over 45 years old, followed in Tabacology unit at CHRU of BREST - No COPD patient or COPD patients not followed for more than 3 years (considered out of care)
* No opposition filed

Exclusion Criteria:

* Patients already followed for COPD
* Contraindication to spirometry
* Refusal to participate

Min Age: 45 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients followed in tabacology unit
Sampling Method: Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2021-05-16 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
COPD DIAGNOSIS | day 1
  The diagnosis of COPD is performed using a spirometry

CONTACTS AND LOCATIONS:
Overall Officials: Marc Beaumont, PhD, Principal Investigator — CH des pays de Morlaix
Locations (1):
- Chu Brest, Brest, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chapman KR, Mannino DM, Soriano JB, Vermeire PA, Buist AS, Thun MJ, Connell C, Jemal A, Lee TA, Miravitlles M, Aldington S, Beasley R. Epidemiology and costs of chronic obstructive pulmonary disease. Eur Respir J. 2006 Jan;27(1):188-207. doi: 10.1183/09031936.06.00024505. No abstract available. PMID 16387952
- [Result] Fuhrman C, Delmas MC; pour le groupe epidemiologie et recherche clinique de la SPLF. [Epidemiology of chronic obstructive pulmonary disease in France]. Rev Mal Respir. 2010 Feb;27(2):160-8. doi: 10.1016/j.rmr.2009.08.003. Epub 2010 Jan 19. French. PMID 20206064